CLINICAL TRIAL: NCT02778321
Title: Prospective Study Evaluating the Interest of Long-term Cardiac Recording in Cerebral Infarction
Acronym: SPIDERFLASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SPIDERFLASH
Record Dates: First submitted 2016-05-09; First posted 2016-05-19 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Neuropathology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Uses of SpiderFlash monitor (Other): The intervention corresponds to the use of Spiderflash as Holter monitor. Investigators will use the SpiderFlash®, Holter monitor (technology "Secure Data") to have a storage capacity enabling a registration up to 30 days with sufficient autonomy.
  A questionnaire evaluating the safety of SpiderFlash® will be given to the patient and the results of Holter will be communicated at the end of the recording to the blinded rhythm specialist.
  Interventions: Device: Uses of SpiderFlash monitor

INTERVENTIONS:
Device: Uses of SpiderFlash monitor — Investigators will use the SpiderFlash®, Holter monitor (technology "Secure Data") to have a storage capacity enabling a registration up to 30 days with sufficient autonomy.
  The data collected :
  * Demographic data: age, sex, vascular risk factors, antithrombotic therapy at the entrance, history of Transient Ischemic Accident (TIA) or Cerebral infarct (CI)
  * Data on the CI:
  * Monitoring Results scope ICU Neurovascular.
  * Presence palpitations
  * Treatment influencing the rate (beta-blockers or antiarrhythmic)
  * Data on cardiac monitoring:
  A questionnaire evaluating the safety of SpiderFlash® will be given to the patient and the results of Holter will be communicated at the end of the recording to the blinded rhythm specialist

SUMMARY:
Cerebral infarction (CI) can be linked to atherosclerosis of large vessels, occlusion of small vessels intracerebral (gaps), a cardioembolic disease or other rare causes. However, up to 40% of CI remains unexplained after a thorough diagnostic workup. They are called cryptogenic IC.

Atrial fibrillation (AF) is the cause of 25% of the CI but it is recognized that episodes of paroxysmal AF, asymptomatic and unnoticed, may be responsible for a portion of the IC cryptogenic pace. Recognition of these episodes is of great importance since they have the same risk embolic the FA continues [1, 2] and motivate anticoagulant therapy startup.

Several recording techniques heart rate were evaluated after the IC for detecting the AF. Their profitability increases with the duration of the recording: about 3% for a typical 24-hour Holter, the AF detection rate increases to 6% for a 7-day surveillance period, to 12-23% for 30 days and 17-26% with implantable recorders long.

Otherwise brief rhythmic heart abnormalities can be detected with the waning of an CI without the significance of these episodes is known.

Investigators decided to conduct this study because there is no prospective study of good quality with a sufficient number of patients that evaluated the interest of a non-invasive recording of long duration. The only randomized CRYSTAL AF is used for invasive subcutaneous implantable monitor (Reveal XT).

To clarify the significance of arrhythmias and because the presence of several causes is common after 65, investigators propose to record all patients hospitalized for HF.

DETAILED DESCRIPTION:
Main objective / secondary The objectives of our study were to assess the prevalence of AF in patients hospitalized for an IC and to detect and describe all heart rhythmic abnormalities reported immediately to the waning of an IC cryptogenic (ie without cause or without obvious cause ) for non-invasive cardiac monitoring.

1. The primary endpoint: number of patients in whom it was found AF
2. Secondary Endpoints: typical patient subgroups in which it was discovered AF and other rhythm abnormalities; Description of the population under prescribed anticoagulation following SpiderFlash® recordings, cardiac ultrasound parameters (including the surface of the left atrium and the index of the function of the mitral annulus) and rhythmic anomalies in groups with atheromatous and cryptogenic stroke.

Inclusion / non inclusion Inclusion criteria

* Patients over 65 years, hospitalized for cerebral infarction ICU Neurovascular
* No history of atrial fibrillation or flutter
* No hypercoagulable
* Patient unopposed and capable of carrying 21-day monitoring Exclusion criteria
* Patients with severe cognitive impairment that can not keep SpiderFlash® for 21 days
* Previous history of AF or flutter
* Significant artery stenosis requiring specific treatment (endarterectomy or stenting)
* FA on arrival at the ICU Neurovascular
* Trucks of a pacemaker or cardiac defibrillator
* Deadline for the IC more than 10 days
* Other sources of cardiac embolism
* Pejorative prognosis (mRS≥5)

The IC is defined as a central focal neurological deficit of sudden onset and is confirmed by a CT scan or MRI.

The minimum workup includes ECG monitoring by continuous cardiac monitoring, transthoracic echocardiography (transesophageal +/-) and a Doppler ultrasound of the supra-aortic trunks and transcranial.

Methodology :

This is an interventional study in routine care, prospective, single-center, blinded for heart rhythm specialist.

Investigators will use the SpiderFlash®, Holter monitor (technology "Secure Data") to have a storage capacity enabling a registration up to 30 days with sufficient autonomy. The SpiderFlash® is currently registered in the GHPSJ for use in various directions including through cryptogenic cerebral infarction.

The data collected will (see Annex 2 CRF):

* Demographic data: age, sex, vascular risk factors, antithrombotic therapy at the entrance, history of Transient Ischemic Accident (TIA) or CI
* Data on the IC: arterial territory, side (right / left) or insular cortex reached severity (NIHSS score) made further examinations, echocardiography result, become during hospitalization (mRS)
* Monitoring Results scope ICU Neurovascular.
* Presence palpitations
* Treatment influencing the rate (beta-blockers or antiarrhythmic)
* Data on cardiac monitoring: time, duration, number of detected events

A questionnaire evaluating the safety of SpiderFlash® will be given to the patient (Appendix 3) and the results of Holter will be communicated at the end of the recording (as will be shown them in the Circular).

During a screening period of one month, 33 eligible patients over 65 admitted to CI 17 patients (51%) were identified including 9 with cryptogenic CI 8 and having either a non-significant atheroma is a rhythm disorder ( ESSV or atrial hyperexcitability). Among 16 ineligible patients, 4 had severe dementia, 11 had previous FA to 1 significant extracranial stenosis.

The patient recruitment period will be one year for one further year or two-year inclusion period to recruit 200 patients originally planned to study (the first year of inclusion has allowed us to include 73 patients) The data will be entered manually on paper CRF and Excel anonymized so not including the patient identifiers (name or IPP).

The originality of our study:

* Prospective study
* Inclusion of CI cryptogenic and non cryptogenic
* Laying SpiderFlash® early after CI
* Correlation with cardiac ultrasound parameters
* Analysis by the blind rhythm specialist (will not be aware of patient characteristics)
* Changing all events while recording (not just the passages FA)
* Questionnaire "comfort" given to the patient

Investigators specify that the data on the comfort of the patient questionnaire will not be transferred to the company Sorin; this questionnaire meets strict medical interest (including estimate the patient's ability to carry equipment during the full period).

Ethics / Regulatory:

The data processing will be carried out locally on the GHPSJ of anonymized way. The inclusion of patients will occur after patient information collection and its non-opposition traced in his medical records (Appendix 1). The data will be entered by the vascular neurologist anonymously. All patient information will remain confidential.

partnerships:

The Sorin company, manufacturer of SpiderFlash® provide (loan) material in sufficient quantity for the duration of the study.

The GHPSJ: neurologist time and CRA The SELARL rythmo: time heart rhythm specialists

ELIGIBILITY:
Inclusion Criteria:

* ICU Neurovascular hospitalized for cerebral infarction CI
* No history of atrial fibrillation or flutter
* No hypercoagulable
* Patient unopposed and capable of carrying 21-day monitoring

Exclusion Criteria:

* Patients with severe cognitive impairment that can not keep SpiderFlash® for 21 days
* Previous history of AF or flutter
* Significant artery stenosis requiring specific treatment (endarterectomy or stenting)
* FA on arrival at the ICU Neurovascular
* Trucks of a pacemaker or cardiac defibrillator
* Deadline for the CI more than 10 days
* Other sources of cardiac embolism
* Pejorative prognosis (mRS≥5)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Cardiac monitoring | During the 30 days of monitoring
  Data concerning cardiac monitoring: time, duration, number of detected events

SECONDARY OUTCOMES:
NIHSS score | Day 1
  Diagnostic and stroke severity score measures the intensity of neurological signs to monitor their progress and estimate their severity.
Treatment influencing the rate | During the 30 days of monitoring
  Treatment influencing the rate (beta blockers or antiarrhythmic drugs)

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu ZUBER, Principal Investigator — Groupe Hospitalier Paris Saint-Joseph (FRANCE)
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France